CLINICAL TRIAL: NCT03295006
Title: A TheraSphere® Advanced Dosimetry Retrospective Global Study Evaluation in Hepatocellular Carcinoma Treatment
Brief Title: A TheraSphere® Advanced Dosimetry Retrospective Global Study in HCC
Acronym: TARGET
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: Biocompatibles UK Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: BTG-007961
Record Dates: First submitted 2017-06-29; First posted 2017-09-27 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: TheraSphere, hepatocellular carcinoma, dosimetry
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Previous Therasphere treatment: Patients who had received TheraSphere yttrium-90 microspheres
  Interventions: Device: TheraSphere

INTERVENTIONS:
Device: TheraSphere — Patients who had received TheraSphere

SUMMARY:
This retrospective, multinational, single-arm study will be conducted in at least 8 sites. An interim analysis will be conducted with data from 100 patients with up to 10 well defined HCC tumor(s) and with at least one tumor ≥3 cm. Normal tissue absorbed dose using pre-procedural 99mTc MAA SPECT or SPECT/CT imaging will be measured to allow the mean absorbed normal tissue dose corresponding to a ≤15% probability of CTCAE grade 3 or higher hyperbilirubinemia (in the absence of disease progression) to be calculated. Total bilirubin will be recorded and graded according to CTCAE version 4.02. All dose-related SAEs at 3 months follow-up will be followed until resolution, death or lost-to-follow-up. AEs related to disease progression will not be considered related to TheraSphere.

DETAILED DESCRIPTION:
Recently published evidence indicates a correlation between yttrium-90 dose delivered to the tumor and normal tissue with safety and efficacy outcomes but there are no validated methods to consistently measure dose delivered to the tumor and normal tissue. In contrast to the standard clinical approach based on average dose to one target volume, this trial, sponsored by Biocompatibles UK, will explore an alternative two-compartment TheraSphere dosimetry methodology to calculate absorbed dose to tumor and normal tissue

ELIGIBILITY:
Inclusion Criteria:

* Up to 10 well defined unilobar/bilobar HCC tumor(s) per lobe with at least one tumor ≥3 cm ± PVT
* Liver dominant disease (limited extra-hepatic metastases in the lung and/or lymph nodes are permitted (up to 5 lesions in the lung, with each individual lesion ≤2cm; any number of lymph node lesions with each individual lesion ≤2 cm).
* Child Pugh stage A or B7.
* BCLC A, B or C.
* Must be male or female, 18 years of age or older.
* Bilirubin ≤2 mg/dL.
* Tumor replacement <50% of total liver volume assessed by diagnostic imaging consisting of multi-phase contrast enhanced CT or contrast enhanced MRI.
* Diagnostic imaging consisting of multi-phase contrast enhanced CT or contrast enhanced MRI within 3 months prior to TheraSphere® administration.
* Infusion of 99mTc-MAA in a single arterial location sufficient to cover up to 10 well-defined tumors per lobe ≤ 6 weeks prior to TheraSphere® administration.
* Patients must have received TheraSphere® in a single treatment setting in one or more arterial locations sufficient to cover up to 10 well-defined tumors based on angiography. Subsequent TheraSphere® treatment to the second lobe may occur at least 4 weeks following the initial TheraSphere® treatment.
* For patients receiving a second TheraSphere® treatment bilirubin levels must have been recorded prior to the second treatment
* Patients must have had clinical evaluation (assessment of liver specific AEs) and laboratory evaluation (at least a serum bilirubin level) at baseline.
* Tumor(s), ≥3 cm, measurable by mRECIST and RECIST 1.1 at baseline

Exclusion Criteria:

* Prior external beam radiation treatment to the liver.
* Prior loco-regional liver directed therapy (cTACE, DEB-TACE and SIR-Spheres).
* Prior liver transplantation.
* Whole liver TheraSphere® treatment following prior liver resection.
* TheraSphere administration to ≤2 segments (e.g., radiation segmentectomy).
* Additional active therapy (TACE and treatment with SIR-Spheres) between first TheraSphere treatment and 3 month (90 days) imaging.
* Hepatic vein invasion.
* Diagnosis of disease progression at peri-procedural imaging as compared to the baseline imaging (physician's discretion).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with up to 10 well-defined unilobar HCC tumors per lobe with at least one tumor ≥3 cm ± PVT.
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2016-10-31 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Alternative two-compartment TheraSphere dosimetry methodology | Baseline
  Normal tissue absorbed dose using pre-procedural 99mTc MAA (Technetium-99m Macroaggregated albumin) SPECT (Single-photon emission computer tomography) or SPECT/CT (Single-photon emission computer tomography/Computer Tomography) imaging, to allow the mean absorbed normal tissue dose corresponding to a ≤15% probability of Common Toxicities Criteria for Adverse Events (CTCAE) grade 3 or higher hyperbilirubinemia (in the absence of disease progression) to be calculated.

SECONDARY OUTCOMES:
Tumor dose | Baseline
  Tumor dose (to tumors ≥3 cm) using pre-procedural 99mTc MAA SPECT or SPECT/CT imaging.
Serious adverse events | 3 months
  All serious adverse events (SAEs) assessed as related or potentially related to TheraSphere
Specific non-serious adverse events (AEs) assessed as related or potentially related to the dose of TheraSphere | 3 months
  Specific non-serious adverse events (AEs) assessed as related or potentially related to the dose of TheraSphere, comprising of any of the following events:
  * Hyperbilirubinemia
  * Ascites
  * Pain
  * Fatigue
  * Nausea
Clinical laboratory assessments | 6 weeks and 3 months
  Clinical laboratory assessments
Objective response (OR) of the target lesion and non-target sesions | 3 months and 6 months
  Objective response (OR) of the target lesion (single largest lesion) and non-target lesion(s) at 3 months and 6 months (if available), and for all scans up to 400 days after TheraSphere administration by Modified Response Evaluation Criteria in Solid Tumors (mRECIST) and Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
Volume changes | 3 and 6 months
  Volume changes (i.e., perfused liver volume and non-perfused liver volume) from baseline afterTheraSphere administration.
Overall Survival (OS) | 6 months
  Overall Survival (OS)
Target Alpha fetoprotein (AFP) response | 6 weeks and 3 months
  Target Alpha fetoprotein (AFP) response (defined as a ≥50% decrease in AFP levels for patients with a baseline AFP level of
  ≥200 ng/mL).
Albumin-bilirubin (ALBI) score | 6 weeks and 3 months
  Albumin-bilirubin (ALBI) score, a measure of liver function for HCC patients after TheraSphere administration.
Dose to Portal Vein Thrombosis (PVT) | baseline, 90 days, 180 days
  Dose to Portal Vein Thrombosis (PVT) based upon pre- and postprocedure imaging (if PVT present).
Dosimetric analysis time | baseline
  Dosimetric analysis time (i.e., workflow).
Dose accuracy | baseline
  Dose accuracy based upon phantom imaging studies.
Dose reproducibility | baseline
  Measurement of inter-observer agreement based on a round robin review of the same 20 patients obtained from a minimum of 8 users (with each user at a different site) and an exploratory assessment of intra-observer agreement based on a review of 10 patients by a minimum of 8 users at least 2 weeks apart. The 10 patients for the intra-observer agreement will be a subset of the patients included in the assessment of inter-observer agreement.

OTHER OUTCOMES:
Normal tissue dose and tumor dose using post-procedural PET/CT Imaging | baseline
  Normal tissue dose and tumor dose (in tumors ≥3 cm) using post-procedural yttrium-90 Positron Emission Tomography/Computed Tomography (PET/CT) imaging; collection of these endpoints will allow an assessment of the correlation with the dose determined from preprocedural 99mTc MAA SPECT or SPECT/CT imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Marnix Lam, MD, PhD, Principal Investigator — Universitair Medisch Centrum Utrecht; Riad Salem, MD, Principal Investigator — Northwestern University; Etienne Garin, MD, Principal Investigator — Centre Eugène Marquis; Hugo de Jong, PhD, Principal Investigator — Universitair Medisch Centrum Utrecht
Locations (14):
- United States (6):
  - Stanford University Medical Center, Stanford, California
  - University of Florida College of Medicine, Gainesville, Florida
  - Northwestern Memorial Hospital, Robert H Lurie Comprehensive Cancer Center, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Washington University in St. Louis, School of Medicine, Saint Louis, Louisiana
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Centre Eugene Marquis, Rennes, France
- Universitätsklinikum Essen, Essen, Germany
- Foundation IRCCS Istituto Nazionale Tumori, Milan, Italy
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands
- King Faisal Hospital, Riyāḑ, Saudi Arabia
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland
- Turkey (Türkiye) (2):
  - Istanbul university Istanbul medical school, Fatih
  - Florence Nightingale, Şişli

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lam M, Garin E, Haste P, Denys A, Geller B, Kappadath SC, Turkmen C, Sze DY, Alsuhaibani HS, Herrmann K, Maccauro M, Cantasdemir M, Dreher M, Fowers KD, Gates V, Salem R. Utility of pre-procedural [99mTc]TcMAA SPECT/CT Multicompartment Dosimetry for Treatment Planning of 90Y Glass microspheres in patients with Hepatocellular Carcinoma: comparison of anatomic versus [99mTc]TcMAA-based Segmentation. Eur J Nucl Med Mol Imaging. 2025 Jan;52(2):744-755. doi: 10.1007/s00259-024-06920-6. Epub 2024 Sep 27. PMID 39331131
- [Derived] Lam M, Garin E, Palard-Novello X, Mahvash A, Kappadath C, Haste P, Tann M, Herrmann K, Barbato F, Geller B, Schaefer N, Denys A, Dreher M, Fowers KD, Gates V, Salem R. Direct comparison and reproducibility of two segmentation methods for multicompartment dosimetry: round robin study on radioembolization treatment planning in hepatocellular carcinoma. Eur J Nucl Med Mol Imaging. 2023 Dec;51(1):245-257. doi: 10.1007/s00259-023-06416-9. Epub 2023 Sep 12. PMID 37698645
- [Derived] Lam M, Garin E, Maccauro M, Kappadath SC, Sze DY, Turkmen C, Cantasdemir M, Haste P, Herrmann K, Alsuhaibani HS, Dreher M, Fowers KD, Salem R. A global evaluation of advanced dosimetry in transarterial radioembolization of hepatocellular carcinoma with Yttrium-90: the TARGET study. Eur J Nucl Med Mol Imaging. 2022 Aug;49(10):3340-3352. doi: 10.1007/s00259-022-05774-0. Epub 2022 Apr 8. PMID 35394152